CLINICAL TRIAL: NCT05192772
Title: EASY CARE Early Neurological Assessment With Pupillometry in Cardiac Arrest During Resuscitation
Brief Title: Early Neurological Assessment With Pupillometry in Cardiac Arrest During Resuscitation
Acronym: EASY-CARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Collaborators: AREU - Agenzia Regionale Emergenza Urgenza (Unknown)
Responsible Party: Principal Investigator, Simone Maria Zerbi, Principal Investigator, Azienda Ospedaliera Sant'Anna
Other Study IDs: 2494
Record Dates: First submitted 2021-11-25; First posted 2022-01-14 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: NPi200 — Digital pupillometry performed during cardiopulmonary resuscutation (CPR) every CPR cycle end in case of not intubated patient, or every 2 minutes in case of intubated patient

SUMMARY:
Easy Care study wants to demonstrate a correlation between intra-CPR infrared quantitative pupillometry and return of spontaneous circulation (ROSC).

Neurological pupil index (NPi) will be used alone and in association with end-tidal CO2.

DETAILED DESCRIPTION:
At the arrival of medicalised rescue team on the emergency scene, patient will be screened for including criteria. In case of eligibility pupillometry will be collected each eye in the following frame time:

* T 0: time of enrolling
* T 1: after first cycle of resuscitation (approximatively 2 minutes following guidelines)
* T 2 … Tn: every cycle of CPR (or every 2 minutes if intubated patient) bilateral pupillometry will be collected
* T end: the last pupillometry at ROSC time or death. All pupillometry mesures will be obtained from a technician not trained to interpret NPi index. This to maintain blindness during resuscitation efforts.

Data will be collected in anonymous web-based database passwords protected. For the survivors patients enrolled, data collecting continue in Intensive Care Unit (ICU) as neuroprognostication exams (biomarkers, imaging, neurophysiology). Blind follow up will be obtained from ICU as described in secondary outcome section

ELIGIBILITY:
Inclusion Criteria:

* Not traumatic cardiac arrest in pre-hospital setting (OHCA)
* unexpected OHCA
* Lombardy region territory

Exclusion Criteria:

* Traumatic Brain injury
* Cerebrovascular emergecies at computer tomography (CT) scan after hospital admission
* Peripheral or cortical blindness
* One or both eyes loss
* Iris palsy or known peripheral anisocoria
* No indication for resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults present in the Lombardy region at the time of cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) prediction | Variable because depends on the cardiac resuscitation manoeuvers lasting usually not more than 45 minutes
  We are searching for possible correlation between pupillary reactivity (NPi) collected during resuscitation manoeuvres and ROSC. NPi is a numeric score ranges from 0 (unreactive pupils) and 5 (normal reflex).

SECONDARY OUTCOMES:
Correlation of NPi and end tidal CO2 (ETCO2) and ROSC prediction | Variable because depends on the cardiac resuscitation manoeuvers lasting usually not more than 45 minutes
  NPi meaning has been described previously, ETCO2 represents the amount of CO2 exhaled during ventilation in course of cardiopulmonary resuscitation. It represent a good indicator of tissues reperfusion.
  We suppose that NPi could reflect the brainstem vitality. We want to demonstrate if the association between a well known indicator as ETCO2 and the NPi may emprove the ROSC prediction compared to NPi alone (primary objective).
Correlation between NPi and Neurological Outcome as Modified Rankin Scale (mRS) | 1 month, 6 months, 1 year
  association between pupillary reactivity (NPi) absence and poor neurological outcome. The outcome will be evaluated in using modified Rankin Scale range from 0 (no symptoms) to 6 (death). We will aggregate the outcome in a dichotomised result as: good outcome (mRS 0-4) and poor outcome (mRS 5-6).
  The exams of patients will be performed at 1 month, 6 month (or hospital discharge) and 1 year from ROSC, and at ICU discharge.
  The patients exams will be performed with a telephone interview about their fisical condition accordingly to mRS score description.
Correlation between NPi trend and ROSC | Variable because depends on the cardiac resuscitation manoeuvers lasting usually not more than 45 minutes
  We are searching for a possible correlation between the NPi trend during cardiac pulmonary resuscitation (CPR) and the ROSC. We suppose that an improvement of NPi values during CPR can indicate a progressive oxygenation and functionality of tissues with an increased probability of ROSC
Correlation between NPi trend and mRS in ROSC patients | 1 month, 6 months, 1 year
  Similarly to outcome 4, we suppose that a progressive improvement of NPi values during CPR may suggest vitality of the brainstem and oxigenation of the brain.
  We want to evaluate possible correlation between changing in NPi trend and neurological outcome with mRS in the survivors patient (ROSC)

CONTACTS AND LOCATIONS:
Overall Officials: Simone M Zerbi, MD, Principal Investigator — ASST Lariana Ospedale Sant'Anna di Como; Frank A Rasulo, Prof., Study Director — Division of Anesthesiology, Intensive Care & emergency Medicine, Università degli studi di Brescia; Marco Botteri, MD, Study Chair — AREU - Agenzia Regionale Emergenza Urgenza; Claudio Sandroni, Prof., Study Chair — Institute of Anesthesiology and Intensive Care Medicine, Università Cattolica del Sacro Cuore, Roma.; Giovanni Chiarini, MD, Study Chair — Dip. Anestesia, Rianimazione ed Emergenze II, ASST Spedali Civili di Brescia; Maurizio Raimondi, MD, Study Chair — UOC Anestesia e Rianimazione Voghera e Oltrepò, ASST Pavia.; Antonio Bellasi, phD, Study Chair — Department of Medicine, Division of Nephrology, EOC, Lugano
Locations (1):
- Agenzia Regionale Emergenza Urgenza - AREU, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oddo M, Sandroni C, Citerio G, Miroz JP, Horn J, Rundgren M, Cariou A, Payen JF, Storm C, Stammet P, Taccone FS. Quantitative versus standard pupillary light reflex for early prognostication in comatose cardiac arrest patients: an international prospective multicenter double-blinded study. Intensive Care Med. 2018 Dec;44(12):2102-2111. doi: 10.1007/s00134-018-5448-6. Epub 2018 Nov 26. PMID 30478620
- [Background] Riker RR, Sawyer ME, Fischman VG, May T, Lord C, Eldridge A, Seder DB. Neurological Pupil Index and Pupillary Light Reflex by Pupillometry Predict Outcome Early After Cardiac Arrest. Neurocrit Care. 2020 Feb;32(1):152-161. doi: 10.1007/s12028-019-00717-4. PMID 31069659
- [Background] Achamallah N, Fried J, Love R, Matusov Y, Sharma R. Pupillary Light Reflex Is Not Abolished by Epinephrine and Atropine Given During Advanced Cardiac Life Support in Patients Who Achieve Return of Spontaneous Circulation. J Intensive Care Med. 2021 Apr;36(4):459-465. doi: 10.1177/0885066620906802. Epub 2020 Feb 18. PMID 32066312
- [Background] Lee HJ, Shin J, Hong KJ, Jung JH, Lee SJ, Jung E, You KM, Kim TH. A feasibility study for the continuous measurement of pupillary response using the pupillography during CPR in out-of-hospital cardiac arrest patients. Resuscitation. 2019 Feb;135:80-87. doi: 10.1016/j.resuscitation.2018.11.016. Epub 2018 Dec 30. PMID 30599180
- [Derived] Zerbi SM, Sandroni C, Botteri M, Bellasi A, Latronico N, Rasulo F. Early Neurological ASsessment with pupillometrY during Cardiac Arrest REsuscitation (EASY-CARE): protocol for an observational multicentre prospective study. BMJ Open. 2022 Dec 20;12(12):e063633. doi: 10.1136/bmjopen-2022-063633. PMID 36600432